CLINICAL TRIAL: NCT06779513
Title: Validation and Assessment of Novel Morphology-Voltage-P-wave Score for Diagnosing Left Ventricular Diastolic Dysfunction in Patients With Hypertension
Acronym: VANESSA
Status: Recruiting | Type: Observational
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Sodiqur Rifqi, Principal Investigator; Former of Head of Department of Cardiovascular Medicine Faculty of Medicine Universitas Diponegoro, Universitas Diponegoro
Other Study IDs: Undip_Kardio 4
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with LVDD: Investigators will assess MVP score by reviewing patient 12-lead ECG. Furthermore, the MVP score will be analyzed with echocardiography result.
  Interventions: Diagnostic Test: Echocardiohraphy
- Patient without LVDD: Investigators will assess MVP score by reviewing patient 12-lead ECG. Furthermore, the MVP score will be analyzed with echocardiography result.
  Interventions: Diagnostic Test: Echocardiohraphy

INTERVENTIONS:
Diagnostic Test: Echocardiohraphy — Transthoracal echocardiography for diastolic function assessment

SUMMARY:
This study aimed to assess and validate the diagnostic utility of a novel Morphology-Voltage-P-wave Score (MVP Score) in identifying left ventricular diastolic dysfunction among patients with hypertension.

Researchers will collect information of patient with hypertension and underwent transthoracal echocardiography assessment. The data consist of demographic data, clinical presentation, laboratory, and echocardiography result were collected by two investigators. Then, the data was analyzed by using IBM SPSS Statistics v26.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension

Exclusion Criteria:

* Secondary or resistant hypertension
* LVEF<55%
* Congenital heart disease
* Infiltrative cardiomyopathy
* Coronary artery disease
* Chronic kidney disease
* Valvular heart disease
* Bundle branch block
* Arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with essential hypertension who came to out hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Diastolic Dysfunction | Up to 1 weeks
  Diastolic Dysfunction found in transthoracal echocardiography assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No